CLINICAL TRIAL: NCT04295655
Title: Feasibility and Efficacy of Physiotherapy in Hypoxic AECOPD Patients
Brief Title: Physiotherapy in Hypoxic AECOPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0089UG
Record Dates: First submitted 2020-02-17; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Global Exercise Group (Experimental): all patients received the Control Group treatment added to global exercise treatment. The program included 15 minutes of deep breathing exercises and 20-30 minutes of limb exercises. The exercises included global active range of motion (ROM) exercises and muscle strengthening like upper and lower limbs flexion-extension do single-leg stance, and sit to stand exercises. The number of repetitions was adapted to the subject's response taken into account the perceived dyspnea and fatigue during the exercise performance.
  Interventions: Other: Global Exercise intervention
- Functional Electrostimulation Group (Experimental): all patients received the Control Group treatment plus neuromuscular stimulation therapy (SEFAR Rehab X2, DJO France S.A.S., France) on quadriceps accompanied by lower limb exercises. The intervention was performed following the protocol described by Valenza et al (2017).
  Valenza MC, Torres-Sánchez I, López-López L, Cabrera-Martos I, Ortiz-Rubio A, Valenza-Demet G. Effects of home-based neuromuscular electrical stimulation in severe chronic obstructive pulmonary disease patients: a randomized controlled clinical trial. Eur J Phys Rehabil Med. 2018 Jun;54(3):323-332. doi: 10.23736/S1973-9087.17.04745-1. Epub 2017 Nov 16. PubMed PMID: 29144103.
  Interventions: Other: Functional Electrostimulation Group
- Standard treatment (Active Comparator): Patients received standard medical and pharmacological care that consisted in systemic steroids, inhaled bronchodilators, oxygen, and a regimen of oral prednisone or its equivalent in doses of 40 to 60 mg per day for the duration of therapy as well as anti-biotic therapy.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Global Exercise intervention — The program included 15 minutes of deep breathing exercises and 20-30 minutes of limb exercises. The exercises included global active range of motion (ROM) exercises and muscle strengthening like upper and lower limbs flexion-extension do single-leg stance, and sit to stand exercises
  Arms: Global Exercise Group
Other: Functional Electrostimulation Group — The program included a neuromuscular stimulation therapy on quadriceps accompanied by lower limb exercises. The intervention was performed following the protocol described by Valenza et al (2017).
  Valenza MC, Torres-Sánchez I, López-López L, Cabrera-Martos I, Ortiz-Rubio A, Valenza-Demet G. Effects of home-based neuromuscular electrical stimulation in severe chronic obstructive pulmonary disease patients: a randomized controlled clinical trial. Eur J Phys Rehabil Med. 2018 Jun;54(3):323-332. doi: 10.23736/S1973-9087.17.04745-1. Epub 2017 Nov 16. PubMed PMID: 29144103.
  Arms: Functional Electrostimulation Group
Other: Standard treatment — Patients received standard medical and pharmacological care that consisted in systemic steroids, inhaled bronchodilators, oxygen, and a regimen of oral prednisone or its equivalent in doses of 40 to 60 mg per day for the duration of therapy as well as anti-biotic therapy
  Arms: Standard treatment

SUMMARY:
Hypoxia is considered a key player in many of the comorbidities that characterize COPD, such as pulmonary hypertension, skeletal muscle dysfunction, and systemic inflammation. These comorbidities are worsened during an exacerbation due to prolonged bed rest and treatment with steroids, showing a reduction in the quality of life, exercise tolerance, and a greater risk of death in these patients. Therefore, a better understanding of the safety and effectiveness of exercise training for AECOPD patients with resting hypoxemia is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* A diagnosis of COPD made according to the criteria of the American Thoracic Society (ATS)
* With hypoxemia at rest defined as mean arterial oxygen saturation below 90%
* Agreed to participate

Exclusion Criteria:

* Unstable cardiovascular disease
* Orthopedic diseases in the upper and lower limbs
* Being in ICU or use of mechanical ventilation
* Motor sequelae from a neurological or cognitive impairment that interfere with the evaluation and the treatment
* Contraindications of electrotherapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Lower limb strength | Baseline
  Quadriceps strength was assessed with a portable hand-held dynamometer (Lafayette Manual Muscle Testing System, model 01163, Lafayette, IN, USA). The test was performed with the patient seated with his/her knees and hips flexed at 90°. Resistance was applied to the anterior tibia during 5 seconds of maximal muscle contraction. The test was repeated alternatively 3 times on the leg, allowing participants to rest between measurements. The highest value in Newton was selected for the analysis.
Lower limb strength | Up to 9 days
  Quadriceps strength was assessed with a portable hand-held dynamometer (Lafayette Manual Muscle Testing System, model 01163, Lafayette, IN, USA). The test was performed with the patient seated with his/her knees and hips flexed at 90°. Resistance was applied to the anterior tibia during 5 seconds of maximal muscle contraction. The test was repeated alternatively 3 times on the leg, allowing participants to rest between measurements. The highest value in Newton was selected for the analysis.
Balance | Baseline
  Balance was evaluated by the one-leg standing balance test (OLS), that measured the time that the patient balances on one leg as long as possible. The patient choose a leg to stand on (whichever he felt more comfortable with), flex the opposite knee allowing the foot to clear the floor, and balance on one leg. Higher values mean better balance.
Balance | Up to 9 days
  Balance was evaluated by the one-leg standing balance test (OLS), that measured the time that the patient balances on one leg as long as possible. The patient choose a leg to stand on (whichever he felt more comfortable with), flex the opposite knee allowing the foot to clear the floor, and balance on one leg. Higher values mean better balance.
Dyspnea | Baseline
  Dyspnea was assessed at rest using the modified Borg scale. Patients classified their breathlessness from 0 (no dyspnea) to10 (maximal dyspnea)
Dyspnea | Up to 9 days
  Dyspnea was assessed at rest using the modified Borg scale. Patients classified their breathlessness from 0 (no dyspnea) to10 (maximal dyspnea)
Fatigue | Baseline
  Fatigue was evaluated using the Piper Fatigue Scale (PFS) that consists of 22 numerical items which assess multidimensional aspects of fatigue. The scale measures four dimensions of subjective fatigue: "behavioral/severity", relating to the severity, distress, and degree of disruption in activity of daily living; "affective meaning", relating to the emotional meaning attributed to fatigue; "sensory", relating to the physical symptoms of fatigue; and "cognitive/mood", relating to mental and mood states
Fatigue | Up to 9 days
  Fatigue was evaluated using the Piper Fatigue Scale (PFS) that consists of 22 numerical items which assess multidimensional aspects of fatigue. The scale measures four dimensions of subjective fatigue: "behavioral/severity", relating to the severity, distress, and degree of disruption in activity of daily living; "affective meaning", relating to the emotional meaning attributed to fatigue; "sensory", relating to the physical symptoms of fatigue; and "cognitive/mood", relating to mental and mood states

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain